CLINICAL TRIAL: NCT02499627
Title: A Phase II Study With Bendamustine Plus Brentuximab Vedotin in Hodgkin's Lymphoma and CD30+ Peripheral T-cell Lymphoma in First Salvage Setting: the BBV Regimen.
Brief Title: Bendamustine Plus Brentuximab Vedotin in HL and CD30+ PTCL in First Salvage Setting
Acronym: FIL-BBV
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: expected accrual not reached
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIL-BBV
Record Dates: First submitted 2015-07-14; First posted 2015-07-16 (Estimated); Last update posted 2021-05-27 (Actual); Status verified 2020-09

CONDITIONS: Lymphatic Diseases
Keywords: Lymphoma; Hodgkin; PTCL; CD30+
MeSH Terms: conditions — Lymphatic Diseases; Lymphoma | interventions — Brentuximab Vedotin; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bendamustine + Brentuximab for 6 cycles (Experimental): Bendamustine 90 mg/m2 d1-2. Brentuximab vedotin 1.8 mg/kg d1.Every 21 days for 6 cycles.
  Interventions: Drug: Brentuximab Vedotin; Drug: Bendamustine

INTERVENTIONS:
Drug: Brentuximab Vedotin — Brentuximab will be given intravenously at a total dose of 1.8 mg/kg on day 1 of each 21 days-based cycle, for 6 cycles.
  Other Names: SGN35
Drug: Bendamustine — Bendamustine will be administered at a dose of 90 mg/m2 on day 1 and 2 of each 21 days-based cycle, for 6 cycles.
  Other Names: Levact

SUMMARY:
This is a single-arm, open-label, multicenter, phase 2 clinical trial aimed at evaluating the efficacy and safety of the combination of bendamustine and brentuximab vedotin as a first salvage therapy in patients with relapsed or refractory Hodgkin's lymphoma or PTCL.

A total of 25 patients with PTCL, and 40 with Hodgkin's lymphoma are expected to be treated according to this treatment protocol.

DETAILED DESCRIPTION:
In the study, intravenous bendamustine will be administered at a dose of 90 mg/m2 on day 1 and 2 and brentuximab will be given intravenously at a total dose of 1.8 mg/kg on day 1 of each 21 days-based cycle, for 6 cycles. All patients achieving a CR can be considered eligible to peripheral blood stem cell mobilization (to be performed with granulocytecolony stimulating factor alone) and may proceed to an ASCT at any time after cycle 4.

ELIGIBILITY:
Inclusion criteria for patients with classical Hodgkin's lymphoma:

1. Patients with primary refractory disease after one previous line of therapy or at first relapse after one previous line of therapy. Patients must have completed any prior treatment with radiation, chemotherapy, biologics, immunotherapy and/or other investigational agents at least 4 weeks prior to the first BBV dose
2. Histologically-confirmed CD30+ disease (IHC BerH2 antibody)
3. Age from 18 to 60 years.
4. Fluorodeoxyglucose (FDG)-avid and measurable disease (lymph nodes must have long axis of 1.5 cm regardless of short axis or long axis 1.1 to 1.5 and short axis > 1.0 cm) as documented by both PET and CT.
5. An Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. The following required baseline laboratory data: absolute neutrophil count (ANC) ≥ 1500/μL, unless known marrow involvement due to disease, platelets ≥ 75,000/μL, unless known marrow involvement due to disease, bilirubin ≤ 1.5 x upper limit of normal (ULN) or ≤ 3 x ULN for patients with Gilbert's disease, serum creatinine ≤ 1.5 X ULN, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 X ULN.
7. Serum Albumin ≥ 3 g/dL.
8. Females of childbearing potential must have a negative serum or urine β-hCG pregnancy test result within 7 days prior to the first dose of therapy. Females of non-childbearing potential are those who are postmenopausal for more than 1 year or who have had a bilateral tubal ligation or hysterectomy.
9. Both females of childbearing potential and males who have partners of childbearing potential must agree to use an effective contraceptive method during the study and for at least 6 months following the last dose of study drug.
10. Male patients, even if surgically sterilized (i.e., post vasectomy), who:

    1. Agree to practice effective barrier contraception during the entire study treatment period and through 6 months after the last dose of the study drug, or
    2. Agree to completely abstain from heterosexual intercourse.
11. Patients must provide written informed consent

Exclusion criteria for patients with classical Hodgkin's lymphoma:

1. Previous treatment with bendamustine or brentuximab vedotin.
2. Prior autologous stem cell transplant.
3. Known history of any of the following cardiovascular conditions: myocardial infarction within 2 years of study entry; NYHA class III or IV heart failure; cardiac arrhythmias; angina; any electrocardiographic evidence of acute ischemia or conduction system abnormalities; recent evidence (within 6 months before the first dose of study drug) of a left-ventricular ejection fraction < 50%.
4. History of another primary malignancy for within 3 years of study entry (the following are exempt from the 3-year limit: non-melanoma skin cancer, curatively treated localized prostate cancer and cervical carcinoma in situ on biopsy or a squamous intraepithelial lesion on PAP smear).
5. Known cerebral/meningeal disease (HL or any other etiology) or testicular involvement.
6. Signs or symptoms of progressive multifocal leukoencephalopathy (PML).
7. Pre-existing Peripheral Neuropathy ≥ 2.
8. Any active systemic viral, bacterial, or fungal infection requiring treatment with antimicrobial therapy within 2 weeks prior to the first dose of therapy.
9. Current therapy with other systemic anti-neoplastic or investigational agents.
10. Therapy with corticosteroids at greater than or equal to 20 mg/day prednisone equivalent within 1 week prior to the first dose of therapy.
11. Women who are pregnant or breastfeeding.
12. Patients with a known hypersensitivity to recombinant proteins, murine proteins, or any excipient contained in the drug formulation of brentuximab vedotin and to bendamustine.
13. HIV positive.
14. HCV positive.
15. HBsAg positive; HBsAg negative patients with anti-HBcAg positive can be enrolled if HBV DNA is negative and antiviral treatment with Lamivudine or Tenofir is provided.
16. Active varicella zoster virus (VZV) infection; previously infected patients is accepted only with concomitant treatment with Valacyclovir or Acyclovir.
17. Patients with dementia or altered mental state that would preclude the understanding and rendering of informed consent.

Inclusion criteria for patients with peripheral T-cell lymphomas:

1. Patients with refractory or relapsed PTCL regardless of the number of prior therapy lines. Patients must have completed any prior treatment with radiation, chemotherapy, biologics, immunotherapy and/or other investigational agents at least 4 weeks prior to the first dose of therapy.
2. Signed written informed consent.
3. Age from 18 to 60 years.
4. Histologically confirmed diagnosis of PTCL, i.e. PTCL-not otherwise specified (PTCL-NOS), angioimmunoblastic T cell lymphoma (AITL) and transformed mycosis fungoides according to the World Health Organization (WHO) 2008 classification.
5. Histologically confirmed CD30+ PTCL (IHC BerH2 antibody).
6. Eastern Cooperative Oncology Group (ECOG) performance status score of ≤ 1 at study entry.
7. At least one site of measurable disease in two dimensions by computed tomography. Both nodal and extranodal sites will be taken into consideration (lymph nodes must have long axis of 1.5 cm regardless of short axis or long axis 1.1 to 1.5 cm and short axis > 1.0 cm).
8. Hematology values within the following limits:

   1. absolute neutrophil count (ANC) ≥ 1500/mm3 independent of growth factor support;
   2. platelets ≥ 75,000/mm3 or ≥ 50,000/mm3 if bone marrow involvement is independent of transfusion support;
   3. hemoglobin level ≥ 8 g/dL.
9. Biochemical values within the following limits:

   1. alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 3 x upper limit of normal (ULN);
   2. total bilirubin < 1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or has a non-hepatic origin);
   3. serum creatinine ≤ 2 x ULN;
   4. serum albumin ≥ 3 g/dL.
10. Women of childbearing potential must have a negative pregnancy test within 7 days of receiving study medication and must agree to use effective contraception, defined as: oral contraceptives, double barrier method or practice true abstinence from sexual intercourse during the study and for at least 6 months after the last dose of study drug.
11. Male subjects and their female partners of childbearing potential must be willing to use an appropriate method of contraception or practice true abstinence from sexual intercourse during the study and for at least 6 months after the last dose of study drug.

Exclusion criteria for patients with peripheral T-cell lymphomas:

1. Diagnosis of cutaneous T-cell lymphoma, anaplastic large-cell lymphoma (ALCL), mycosis fungoides or Sézary Syndrome.
2. Previous treatment with bendamustine or brentuximab vedotin.
3. Known hypersensitivity to recombinant proteins, murine proteins, or to any excipient contained in the drug formulation of brentuximab vedotin and to bendamustine.
4. Any serious active disease or co-morbid medical condition (according to investigator's decision).
5. Prior history of malignancies other than lymphoma (except for a history of a complete resection for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast) unless the subject has been free of the disease for ≥ 3 years.
6. Pre-existing peripheral neuropathy grade ≥ 2.
7. Signs or symptoms of progressive multifocal leukoencephalopathy (PML).
8. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
9. Pregnant or lactating females or men or women of childbearing potential not willing to use an adequate method of birth control for the duration of the study or a positive pregnancy test on day 1 before first dose of study drug.
10. Central nervous system disease (meningeal and/or brain involvement by lymphoma) or testicular involvement.
11. History of clinically relevant liver or renal insufficiency; significant pulmonary, gastrointestinal, endocrine, neurologic, rheumatologic, hematologic, psychiatric, or metabolic disturbances.
12. Known history of any of the following cardiovascular conditions: myocardial infarction within 2 years of study entry; NYHA class III or IV heart failure; cardiac arrhythmias; angina; any electrocardiographic evidence of acute ischemia or conduction system abnormalities; recent evidence (within 6 months before the first dose of study drug) of a left-ventricular ejection fraction < 50%.
13. Active systemic, viral, bacterial, or fungal infection requiring systemic antibiotics within 2 weeks prior to first dose of study drug.
14. HIV positive.
15. HCV positive.
16. HBsAg positive; HBsAg negative patients with anti-HBcAg positive can be enrolled if HBV DNA is negative and antiviral treatment with Lamivudine or Tenofir is provided.
17. Active varicella zoster virus (VZV) infection; previously infected patients is accepted only with concomitant treatment with Valacyclovir or Acyclovir.
18. Prior allogeneic stem cell transplant
19. Patients with dementia or altered mental state that would preclude the understanding and rendering of informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2015-12-23 (Actual); Primary Completion 2019-09-13 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Overall objective response rate (ORR). | 1 year
  Proportion of patients in CR or PR

SECONDARY OUTCOMES:
Duration of the response (DOR) | 1 year
  Time from documentation of tumor response to disease progression
Complete remission (CR) rate | 1 year
  Proportion of patients in CR
Progression-free survival (PFS) | 1 year
  Time from study enrollment until disease progression or death
Adverse Events | 1 year
  The type, incidence, severity, seriousness, of adverse events and laboratory abnormalities observed during treatment and the assessment of any potential relationship to the study drugs.
Overall survival (OS) | 1 year
  Time from study enrollment until death from any cause

OTHER OUTCOMES:
One-year event-free survival (EFS) | 1 year
  Time from study enrollment to disease progression, death, or discontinuation of treatment for any reason (eg, toxicity, patient preference, or initiation of a new treatment without documented progression)
B symptoms resolution rate (when documented at presentation) | 1 year
  Proportion of patients with B symptoms at the end of study
CD30 expression and the objective response | 1 year
  Correlation between the CD30 expression and the objective response obtained

CONTACTS AND LOCATIONS:
Overall Officials: Vittorio Stefoni, MD, Principal Investigator — Ematologia "L. & A. Seragnoli" - Policlinico S. Orsola Malpighi
Locations (5):
- Italy (5):
  - A.O S.Orsola-Malpighi, Bologna, BO
  - Spedali Civili, Brescia, BS
  - Fondazione IRCCS Milano INT, Milan, MI
  - AOU Città della Salute e della Scienza, Torino, TO
  - IRCCS Fondazione Pascale, Napoli